CLINICAL TRIAL: NCT02594033
Title: A Single Centre, Randomised, 3-period Cross-over Trial to Investigate Different Needle Features Assessed by Comparing Insulin Aspart Pharmacokinetic Profiles
Brief Title: A Trial to Investigate Different Needle Features Assessed by Comparing Insulin Aspart Pharmacokinetic Profiles
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: INS-4219; U1111-1164-2873 (Other: WHO)
Record Dates: First submitted 2015-10-30; First posted 2015-11-02 (Estimated); Last update posted 2017-08-01 (Actual); Status verified 2017-07

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus | interventions — Insulin Aspart

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- 3 mm needle (Experimental)
  Interventions: Drug: insulin aspart
- 3.5 mm needle (Experimental)
  Interventions: Drug: insulin aspart
- 4 mm needle (Active Comparator)
  Interventions: Drug: insulin aspart

INTERVENTIONS:
Drug: insulin aspart — All subjects make three intervention visits with at least 5 days between individual intervention visits. At each intervention visit the subject receives one insulin aspart injection with only one type of needle.

SUMMARY:
This trial is conducted in Europe. The aim of the trial is to investigate different needle features assessed by comparing insulin aspart Pharmacokinetics profiles (the exposure of the trial drug in the body)

ELIGIBILITY:
Inclusion Criteria:

* Informed consent obtained before any trial-related activities. Trial-related activities are any procedures that are carried out as part of the trial, including activities to determine suitability for the trial
* Male, age at least 18 years at time of signing informed consent
* Considered generally healthy upon completion of medical history, physical examination, analysis of laboratory safety variables, vital signs and ECG (electrocardiogram), as judged by the investigator
* Body mass index (BMI) 28-39.9 kg/m^2 (overweight to obese)
* Caucasian

Exclusion Criteria:

* Male of reproductive age who or whose partner(s) is not using adequate contraceptive methods (adequate contraceptive measures as required by local regulation or practice)
* Non-fasting blood glucose test with blood glucose values above 11.1 millimol per liter (mmol/L)
* HbA1c (Glycosylated Haemoglobin) equal to or above 6.5%
* Known active or in-active skin disease in the injection area or that could affect pain perception
* History of deep leg vein thrombosis or repeated episodes of deep leg vein thrombosis in 1st degree relatives (parents, siblings or children) as judged by the investigator
* Use of any prescription or non-prescription medication, including herbal products and nonroutine vitamins, within the last 2 weeks before screening
* Smoker (defined as a subject who is smoking more than 5 cigarettes or the equivalent per day) who is not able or willing to refrain from smoking or use of nicotine gum or transdermal nicotine patches during the inpatient period
* Known or suspected abuse of alcohol (defined as regular intake of more than 14 units weekly for men where 1 unit equals 300 milliliter (mL) of beer, 100 mL of wine, or 25 mL of distilled spirits)
* Positive result of an alcohol breath test
* Known or suspected drug/chemical substance abuse within 1 year from screening

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2015-10-27 (Actual); Primary Completion 2016-01-28 (Actual); Study Completion 2016-01-28 (Actual)

PRIMARY OUTCOMES:
Area under curve insulin aspart measured in serum | During a maximum of 8 hours
Maximum concentration of insulin aspart measured in serum | During a maximum of 8 hours

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Neuss, Germany

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com